CLINICAL TRIAL: NCT06090955
Title: Modulating Surgery-Induced Blood-Brain Barrier Disruption in Elderly: Impact of Dexmedetomidine and Lidocaine, a Randomized Controlled Trial
Brief Title: Modulating Surgery-Induced Blood-Brain Barrier Disruption in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jiseon Jeong, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SMC 2023-07-162
Record Dates: First submitted 2023-10-03; First posted 2023-10-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Delirium, Postoperative
Keywords: Postoperative delirium; dexmedetomidine; lidocaine; neuroinflammation; CPAR; blood brain barrier
MeSH Terms: conditions — Emergence Delirium; Neuroinflammatory Diseases | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine group (Experimental): Patients in the dexmedetomidine group will be administered a bolus of 0.3 ug/kg intravenous dexmedetomidine over 10 min before anesthetic induction. After bolus injection, a continuous infusion of 0.3 ug/kg/hr of intravenous dexmedetomidine will be administered until the end of surgery.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Lidocaine group (Experimental): Patients in the lidocaine group will receive a bolus of 1.5 mg/kg intravenous lidocaine over 10 min before induction of anesthesia. A continuous infusion of 1.5 mg/kg/hour of systemic lidocaine will be administered until the end of the surgery.
  Interventions: Drug: Lidocaine IV
- Control group (Placebo Comparator): Patients in the control group will be administered equal volumes of 0.9% saline using the identical application scheme.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — The study drugs(dexmedetomidine 80 μg/20 mL) will be prepared with 20 mL syringe and marked as 'trial drug', which are identical in appearance with control and active comparator. In order to avoid anaesthesiologists' speculation about the randomised assignment, the study drugs will be infused at the same rate.
  Other Names: Dex
  Arms: Dexmedetomidine group
Drug: Lidocaine IV — The study drugs(lidocaine 400 mg/20 mL) will be prepared with 20 mL syringe and marked as 'trial drug', which are identical in appearance with control and active comparator. In order to avoid anaesthesiologists' speculation about the randomised assignment, the study drugs will be infused at the same rate.
  Other Names: Lido
  Arms: Lidocaine group
Drug: normal saline — The study drugs(normal saline) will be prepared with 20 mL syringe and marked as 'trial drug', which are identical in appearance with control and active comparator. In order to avoid anaesthesiologists' speculation about the randomised assignment, the study drugs will be infused at the same rate.
  Other Names: Control
  Arms: Control group

SUMMARY:
Postoperative delirium (POD) is the most common complications (~50-60%) in elderly and major challenges to our rapidly growing aging population. Growing evidence suggests a possible role for neuroinflammation in the development of delirium, which is facilitated by a transient increase in blood-brain barrier (BBB) permeability. Lidocaine and dexmedetomidine, commonly used anesthetic adjuncts, have anti-inflammatory properties. Both drugs are reported to have modulatory effect on the intergrity of BBB and associated with a beneficial effect on postoperative neurocognitive dysfunction. In this regard, The investigators aimed to prospectively compare the modulatory effect of the intraoperative administration of dexmedetomidine or lidocaine with a sham control group (normal saline solution) on surgery-induced BBB disruption.

DETAILED DESCRIPTION:
Postoperative delirium (POD) negatively affects cognitive domains including memory, attention, and concentration after surgery. The incidence of POD in high-risk populations, such as aged, patients in intensive care units (ICU) and with previous cognitive impairment, the incidence of POD is as high as 50 to 60%. POD is associated with increased morbidity, mortality, and health-care costs. The 1-year survival probability is reduced by approximately 10% for each additional day of POD. Additionally, it is closely related to long-lasting postoperative cognitive dysfunction.

Surgical trauma activates the innate immune system and central nervous system (CNS) is influenced by surgical trauma by inflammatory mediators rapidly reaching the brain, which is facilitated by a transient increase in blood-brain barrier (BBB) permeability. Recent neuroimaging studies demonstrated BBB dysfunction in patients with delirium after cardiac surgery. The biomakers indicative of BBB breakdown were recently associated with the onset and intensity of delirium. These findings imply that the BBB could serve as a pivotal interface in regulating neuroinflammation and cognitive deterioration following surgical procedures.

Dexmedetomidine and lidocaine are increasingly used as part of a multimodal intraoperative anesthetic adjunct in a variety of surgical procedures. Dexmedetomidine, as a highly selective central presynaptic α2-adrenergic agonist, has sedative, sympatholytic and anti-inflammatory effects. Perioperative dexmedetomidine administration reduced delirium incidence by up to 50% and duration by 0.7 days in surgical populations. Lidocaine, an amide local anesthetic and class-1 antiarrhythmic agent, also has anti-inflammatory and opiate-sparing effects, accelerating gastrointestinal recovery and reducing hospital length of stay. In addition, previous clinical researches have suggested a beneficial effect of perioperative systemic lidocaine on postoperative neurocognitive dysfunction. Although both drugs alleviate surgery-induced systemic inflammation and animal models have indicated a potential protective effect of these agents against surgery-induced disruption of the BBB, few studies have examined the role of these different anesthetics in the interplay between peripheral and central inflammation in human subjects.

In this regard, this study aimed to prospectively compare the modulatory effect of the intraoperative administration of dexmedetomidine or lidocaine with a sham control group (normal saline solution) on surgery-induced BBB disruption in a randomized, placebo-controlled, double-blind, triple-parallel clinical trial. The primary outcome measure was "cerebrospinal-plasma albumin ratio (CPAR)", which is a gold standard measure for BBB permeability, presenting in vivo evidence for the physical breakdown of the blood-CSF barrier in human. The investigators hyptothesized that the use of intraoperative continuous infusion of dexmedetomidine or lidocaine would be statistically superior to placebo control in preserving BBB integrity.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status classification I-III
2. Undergoing elective open pancreatoduodenectomy
3. Voluntary participation in the trial and signed informed consent

Exclusion Criteria:

1. Sinus bradycardia (heart rate (HR) <50 beats per minute (bpm)), Adams-Stokes syndrome, sick sinus or Wolff-Parkinson-White syndrome, or second-degree trioventricular block and over.
2. Concurrent treatment with a class 1 antiarrhythmic or amiodarone)
3. History of hypersensitivity reactions or contraindications to the study drugs (dexmedetomidine or lidocaine).
4. Patient at personal of familial risk of malignant hyperthermia and porphyria
5. Body mass index (BMI) ˃40 kg/m2
6. Patients with coagulopathy (INR 1.5 or more, platelet count less than 75000/ul) or other contraindications to spinal tapping, or on anticoagulants that would preclude safe lumbar punctures.
7. History of severe hepatic (Childs-Pugh Score > Class A ) or renal (glomerular filtration rate <30m)/min×1.73m2) disorders.
8. Severe audio-visual impairments, or inability to speak precluding communication.
9. Evidence of preoperative delirium (Confusion Assessment Method, CAM)
10. History of uncontrolled seizures.
11. Patients on immunosuppressants (e.g., steroids) or immunomodulatory therapy, chemotherapeutic agents with known cognitive effects.
12. Patients taking the following drugs that are moderate-strong inhibitors of the CYP1A2 and CYP3A4 metabolic pathways within 72 hours prior to surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative change of cerebrospinal-plasma albumin ratio (CPAR) | From the baseline to immediate postoperative values
  The change of CPAR will be calculated. CPAR was calculated using the formula 1000 x (CSF albumin (mg/dl))/(serum albumin (mg/dl).

SECONDARY OUTCOMES:
The changes of inflammatory biomarker level in blood | From the baseline to immediate postoperative state and postoperative day 2
  IL-6
The changes of neuronal damage biomarker level in blood | From the baseline to immediate postoperative state and postoperative day 2
  neuron specific enolase
The changes of inflammatory, neuronal damage, BBB permeability biomarker level in blood | From the baseline to immediate postoperative state and postoperative day 2
  sb100 protein
The incidence of postoperative delirium | From postoperative day 0 to 5
  Intensive Care Unit (CAM-ICU) and 3-min diagnostic interview for CAM (3D-CAM) for ICU patients and ward patients, respectively
The subtype of postoperative delirium | From postoperative day 0 to 5
  hyperactive, hypoactive or mixed type will be defined by RASS score
Delirium Rating Scale Revised (DRS-R-98) | From postoperative day 0 to 5
  The severity of delirium will be assessed using the Delirium Rating Scale Revised (DRS-R-98)
Onset and duration of delirium | From postoperative day 0 to 5
  Intensive Care Unit (CAM-ICU) and 3-min diagnostic interview for CAM (3D-CAM)
Pain score (NRS) | From postoperative day 0 to 5
  The degree of surgical pain will be assessed at rest, when taking a deep breath, and when moving by NRS.
Subjective sleep quality | From postoperative day 0 to 5
  the NRS (an 11-point scale where 0 = the best sleep, and 10 = the worst sleep) once daily
Montreal cognitive Assessment (MoCA) | at baseline and 7 days after surgery or at discharge
  Cognitive assessment
Ideal outcome of pancreatoduodenectmoy | postoperative day 30
  defined by the absence of In-hospital mortality, Severe complications (Clavien Dindo ≥3), Postoperative pancreatic fistula - ISGPS Grade B/C, Reoperation, Length of stay >75th percentile, or Readmission
non-delirium complications within 30 days after surgery | Within 30 days after surgery
  The severity of non-delirium complications are graded using Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Jiseon Jeong, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Study data may be made available on request to the principal investigators with an appropriate research and data-protection plan agreed on.